CLINICAL TRIAL: NCT00905541
Title: Influence of Simvastatin on apoB-100 Secretion in Non-Obese Subjects With Moderate Hypercholesterolemia: A Stable Isotope Study
Brief Title: Influence of Simvastatin on Apolipoprotein B-100 (apoB-100) Secretion
Acronym: SVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Heiner K. Berthold, MD, PhD, University of Bonn
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SVS0001
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No treatment (No Intervention): Phase A: No treatment
- simvastatin chronic (Experimental): Phase B: 40 mg/day simvastatin
  Interventions: Drug: simvastatin
- simvastatin acute-on-chronic (Experimental): Phase C: 80 mg simvastatin acute-on-chronic
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: simvastatin — 40 mg/day
  Arms: simvastatin chronic
Drug: simvastatin — 80 mg simvastatin acute-on-chronic
  Arms: simvastatin acute-on-chronic

SUMMARY:
3-Hydroxy-3-methylglutaryl coenzyme A-reductase inhibitors (statins) decrease apolipoprotein B-100-containing lipoproteins by increasing their fractional catabolic rates through low-density lipoproteins (LDL) receptor-mediated uptake. Their influence on hepatic secretion of these lipoproteins is controversial. The current study investigates whether simvastatin influences lipoprotein secretion.

DETAILED DESCRIPTION:
3-Hydroxy-3 methylglutaryl (HMG) coenzyme A-reductase inhibitors (statins) have an established role in the treatment of hypercholesterolemia. Their efficacy in reducing cardiovascular morbidity and mortality in secondary and primary prevention has been demonstrated in large prospective trials. HMG-CoA-reductase inhibitors inhibit competitively the rate-limiting enzyme of endogenous cholesterol biosynthesis. As a consequence, the intracellular pool of free cholesterol decreases and low-density lipoprotein (LDL) receptors are up-regulated, leading to an increased receptor-mediated clearance of LDL from plasma. This mechanism is responsible for a large proportion of their cholesterol-lowering effect. However, a statin-induced decrease in lipoprotein production has also been proposed as a mechanism for their lipid-lowering effects. The underlying mechanisms in vivo, however, that would mediate such an effect, are not fully understood. Except for their pronounced cholesterol-lowering properties, statins have also a modest effect (about 15 to 20%) in decreasing triglyceride concentrations. In subjects with high intra-abdominal fat stores, an increased flux of free fatty acids to the liver produces an increased rate of hepatic triglyceride synthesis, which in turn leads to increased very low-density lipoprotein (VLDL) production, since the latter is partly determined by the intracellular availability of triglycerides. This is also found in subjects with type 2 diabetes mellitus and there are a number of studies showing that in this pathophysiologic state statins are able to decrease lipoprotein production. Interestingly, in obese individuals it has been shown that statins increase the catabolism of apoB-100-containing lipoproteins but do not alter their rates of production or secretion.

In the present study we focus on subjects with near normal body weight (mean body mass index 25 +- 3 kg/m2) and normal serum triglyceride concentrations to investigate, in the fasting state, whether statins influence hepatic lipoprotein production. Since recent evidence suggests that the supply of cholesterol available for incorporation into nascent lipoprotein particles also exerts a regulatory influence on apoB secretion by the liver, we investigate in addition the acute inhibitory effects of a high bolus dose of simvastatin in order to stimulate LDL receptor expression to a maximum degree.

The main goal of the present study is to determine the influence of simvastatin on apoB-100 appearance rates and lipoprotein kinetics in fasting non-obese subjects with moderate hypercholesterolemia. For this purpose, each subject will be investigated with three turnover protocols: once without treatment, once during chronic simvastatin treatment at a standard dosage, and once during chronic simvastatin treatment after an additional acute-on-chronic high bolus dose of simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Hypercholesterolemia

Exclusion Criteria:

* Obesity
* Treatment with lipid-lowering drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1998-11; Primary Completion 1999-03 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
apoB-100 kinetic parameters | One year

SECONDARY OUTCOMES:
Lipoprotein concentrations | One year

CONTACTS AND LOCATIONS:
Overall Officials: Heiner K. Berthold, MD, PhD, Principal Investigator — University of Bonn
Locations (1):
- University of Bonn, Bonn, Germany